CLINICAL TRIAL: NCT06605209
Title: A Prospective, Multi-Center, Non-Randomized, Single-Arm Study Evaluating the Peripheral Balloon-Expandable Covered Stent System for the Treatment of Stenosis and/or Occlusive Lesions in the Common and External Iliac Arteries.
Brief Title: Safety and Effectiveness of the Peripheral Balloon-Expandable Covered Stent System for Iliac Artery Stenosis/Occlusion. (SELECT)
Acronym: SELECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZRD-11
Record Dates: First submitted 2024-09-12; First posted 2024-09-20 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Artery Disease (PAD)
Keywords: Covered Stent; iliac artery
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peripheral Balloon-Expandable Covered Stent System Group (Experimental): This arm of the study involves the use of the Peripheral Balloon-Expandable Covered Stent System. The intervention consists of implanting this stent system into the common and/or external iliac arteries of participants who have been diagnosed with stenosis and/or occlusion. The stent system is designed to be balloon-expandable and covered, providing a means to treat arterial blockages.
  Participants in this arm will undergo the stent implantation procedure, followed by scheduled follow-up visits at discharge, and at 1, 6, 12, 24, and 36 months post-procedure. During these visits, the safety and effectiveness of the stent system will be assessed based on predefined performance goals, including clinical outcomes and any adverse events related to the stent.
  Interventions: Device: Peripheral Balloon-Expandable Covered Stent System

INTERVENTIONS:
Device: Peripheral Balloon-Expandable Covered Stent System — The intervention in this clinical trial involves the Peripheral Balloon-Expandable Covered Stent System. This stent system is specifically designed for the treatment of stenosis and/or occlusion in the common and external iliac arteries.

SUMMARY:
This is a prospective, multi-center, single-arm clinical trial to evaluate the Peripheral Balloon-Expandable Covered Stent System for treating stenosis and/or occlusion in the common and external iliac arteries. The safety and effectiveness of the stent system will be compared to pre-set performance goals. All treated subjects will have follow-up visits at discharge, and at 1, 6, 12, 24, and 36 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 80 years, regardless of sex;
* Participants diagnosed with atherosclerotic disease of the common iliac or external iliac artery;
* Participants with a Rutherford classification of 2 to 4 for the target limb;
* Participants or their legal representatives must be able to understand the study's purpose, demonstrate adequate compliance with the study protocol, and sign the informed consent form.

Exclusion Criteria:

* Pregnant or planning to become pregnant, or breastfeeding women;
* Participants who have previously had a vascular graft implanted in the native iliac artery;
* Participants who have had a stroke or myocardial infarction within 3 months prior to enrollment;
* Participants with known uncorrectable bleeding disorders or severe coagulation abnormalities (PT or APTT ≥ 2 times the upper limit of normal; or platelet count < 80×10^9/L);
* Participants with serum creatinine ≥ 221 μmol/L (2.5 mg/dL) or currently undergoing dialysis;
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2 times the upper limit of normal;
* Severe anemia (hemoglobin level < 60.0 g/L);
* Participants known to be allergic or intolerant to cobalt-based alloys, expanded polytetrafluoroethylene (ePTFE), aspirin, clopidogrel, heparin, rivaroxaban, paclitaxel, contrast agents, or other study materials and medications;
* Participants who have undergone vascular intervention within 30 days prior to surgery or who plan to undergo vascular intervention within 30 days following surgery;
* Participants who have received intra-arterial thrombolysis treatment in the target vessel within 14 days prior to enrollment;
* Participants with significant organ dysfunction or other severe conditions that may lead to non-compliance with the study protocol, affect data interpretation, or have a life expectancy insufficient to complete the clinical trial;
* Participants currently involved in a clinical trial of investigational drugs, biologics, or medical devices;
* Other conditions that, in the investigator's opinion, make the participant unsuitable for the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
primary patency | 12 months
  Primary patency of target lesion at 12-months assessed by duplex ultrasound and adjudicated by an independent core laboratory

SECONDARY OUTCOMES:
Major Adverse Event | 36 months
  Percentage of study subjects experiencing a major adverse event (MAE) defined as: device or procedure-related death, myocardial infarction (MI), target lesion revascularization (TLR) or major amputation of the target limb.
Secondary Patency | 6, 12, 24, and 36 Months
  The secondary patency of target lesion at 6, 12, 24, and 36 Months assessed by duplex ultrasound and adjudicated by an independent core laboratory

CONTACTS AND LOCATIONS:
Locations (1):
- The First Medical Centre, Chinese PLA General Hospital, Beijing, Beijing Municipality, China